CLINICAL TRIAL: NCT03820830
Title: A Phase III Open-label, Multicenter, Randomized Trial of Adjuvant Palbociclib in Combination With Endocrine Therapy Versus Endocrine Therapy Alone for Patients With Hormone Receptor Positive / HER2-negative Resected Isolated Locoregional Recurrence of Breast Cancer
Brief Title: Palbociclib for HR Positive / HER2-negative Isolated Locoregional Recurrence of Breast Cancer
Acronym: POLAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 59-19; 2018-003553-19 (EudraCT Number); BIG 18-02 (Other: Breast International Group (BIG)); WI239003 (Other: Pfizer number)
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Recurrent
Keywords: hormone receptor positive breast cancer; HER2 receptor negative; CDK4/6 inhibitor
MeSH Terms: interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palbociclib plus standard endocrine therapy (Experimental): Palbociclib 125 mg/day tablet taken orally for 21 days, followed by 7 days rest for 3 years from randomization, plus standard endocrine therapy for at least 3 years from randomization.
  Interventions: Drug: Palbociclib 125mg; Drug: Standard endocrine therapy
- Standard endocrine therapy (Active Comparator): Aromatase inhibitor (anastrozole or exemestane or letrozole) oral daily tablet, or Selective Estrogen Receptor Modulator (SERM) such as tamoxifen oral daily tablet or fulvestrant (Faslodex) injection once every 2 weeks for 3 doses then every month. Premenopausal women and men may also receive an LHRH (luteinizing hormone-releasing hormone) agonist by injection. Standard endocrine therapy will be given for at least 3 years from randomization.
  Interventions: Drug: Standard endocrine therapy

INTERVENTIONS:
Drug: Palbociclib 125mg — Palbociclib 125 mg oral tablet taken daily for 3 years from randomization
  Other Names: Ibrance; PD-0332991
  Arms: Palbociclib plus standard endocrine therapy
Drug: Standard endocrine therapy — Aromatase inhibitor (anastrozole or exemestane or letrozole) oral daily tablet, or Selective Estrogen Receptor Modulator (SERM) such as tamoxifen oral daily tablet or fulvestrant (Faslodex) injection once every 2 weeks for 3 doses then every month. Premenopausal women and men may also receive an LHRH (luteinizing hormone-releasing hormone) agonist by injection. Standard endocrine therapy will be given for at least 3 years from randomization.

SUMMARY:
POLAR is a phase III clinical trial, which will test the safety and efficacy of an investigational combination of drugs to learn whether the combination of drugs works for a specific cancer. Palbociclib (Ibrance®) is the name of the investigational agent, which is assessed together with standard anti-hormone therapy in this study. Palbociclib is used to treat patients with hormone receptor-positive / HER2-negative breast cancer which has spread beyond the original tumor and/or to other organs.

During this study, anti-hormone therapy will consist of either a selective estrogen receptor modulator (such as tamoxifen) or an aromatase inhibitor (anastrozole, letrozole, exemestane) or fulvestrant (Faslodex®). Premenopausal women and men may also receive a drug called an LHRH (luteinizing hormone-releasing hormone) agonist by injection.

It is standard of care for people with hormone receptor positive breast cancer to take anti-hormone therapy. The study doctor will determine the type of standard anti-hormone therapy that will be given during this trial.

The purpose of the POLAR study is to compare the effect of using 3 years of palbociclib in combination with standard anti-hormone therapy with standard anti-hormone therapy alone and to evaluate the time until the breast cancer returns, if it does return.

DETAILED DESCRIPTION:
Local or regional recurrence of breast cancer after mastectomy or lumpectomy indicates a poor prognosis, and accompanies or precedes distant metastasis in a high proportion of patients. Patients with isolated locoregional recurrences (ILRR), without evidence of distant metastasis hold a substantial risk of developing subsequent distant metastasis, with 5-year survival probabilities ranging between 45% and 80% after locoregional recurrence. These outcomes show the powerful negative prognostic importance of ILRR events and the need for treatments beyond surgical removal of the ILRR.

Adjuvant chemotherapy and endocrine therapies reduce the risk of relapse and death in patients with primary breast cancer. However, few data are available to inform the recommendation of systemic treatment for locoregional recurrence.

The International Breast Cancer Studies Group carried out the CALOR trial, Chemotherapy as Adjuvant for Locally Recurrent breast cancer (IBCSG 27-02 / BIG 1-02 / NSABP B-37), in collaboration with the Breast International Group (BIG) and the National Surgical Adjuvant Breast and Bowel Project (NSABP), to establish whether chemotherapy improves the outcome of patients with ILRR. An updated, final analysis of CALOR after median follow-up of about 9 years was published in the Journal of Clinical Oncology in April 2018, which confirmed chemotherapy benefitted patients with resected ER-negative ILRR and did not support the use of chemotherapy for ER-positive ILRR.

CALOR results strongly suggest that tailoring treatment according to the disease characteristics of the recurrent lesion, in this case ILRR, provides a better indication of the possible responsiveness to treatment than relying on the characteristics of the primary tumor.

Palbociclib has been granted FDA approval in the U.S. for the treatment of HR-positive/HER2-negative advanced breast cancer in combination with the hormonal treatments letrozole and fulvestrant given the unprecedented results in terms of efficacy of two pivotal clinical trials (PALOMA-2 and PALOMA-3). Palbociclib and other CDK4/6 inhibitors have also shown a good toxicity profile and therefore are ideal candidates for combination with hormonal therapy. CDK4/6 pathway activation is a well-known mechanism of resistance to endocrine therapy, indeed CDK4/6 inhibitors have shown activity in cellular models of acquired resistance to endocrine therapies.

The reason for prolonged duration of palbociclib in the adjuvant setting (2 years) comes from the evidence of preclinical studies where cell senescence was investigated as an appealing mechanism of cell death and was indeed observed in vitro after exposure of breast cancer cells and tumors to a combination of endocrine therapy and palbociclib. It is therefore hypothesized that the longer patients receive combined treatment with palbociclib and an antiestrogen, the more likely they may derive prolonged clinical benefit.

Based on the results of the CALOR trial and on strong evidence of activity of the combination of CDK4/6 inhibitors and endocrine therapy, the hypothesis of the POLAR trial is that the CDK4/6 inhibitor palbociclib in combination with endocrine therapy may be active as adjuvant therapy in patients with HR-positive/HER2-negative resected isolated locoregional recurrence of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer, defined as first proven ipsilateral local and/or regional recurrence of a primary invasive breast cancer in at least one of these sites:

   * breast;
   * the chest wall including mastectomy scar and/or skin;
   * axillary or internal mammary lymph nodes.
2. Completion of locoregional therapy:

   * completion of gross excision of recurrence within 6 months prior to randomization;
   * completion of radiotherapy (if given) more than 2 weeks prior to randomization
3. Negative or microscopically involved margins
4. Female or male aged 18 years or older
5. ECOG performance status 0 or 1
6. Recurrent tumor must be hormone receptor positive: ER+ and/or PgR+ ≥1% by IHC
7. Recurrent tumor must be HER2-negative (0, 1+, 2+ by IHC and/or ISH/FISH not amplified).Tumor with HER2 status 2+ by IHC must also be negative (not amplified) by ISH/FISH

8.-10. Normal hematological, renal, and liver function 11. The patient agrees to make tumor (diagnostic core biopsy or surgical specimen of ipsilateral isolated locoregional recurrence) available for submission for central pathology review 12. Patients must either be planned to initiate, or have already started, endocrine therapy for ipsilateral isolated locoregional recurrence 13.) Written Informed Consent prior to randomization

Exclusion Criteria:

1. Recurrence of any size with direct extension to the chest wall and/or to the skin (ulceration or skin nodules) not surgically removable
2. Evidence of distant metastasis as based on conventional staging examinations (physical, chest X-ray or CT, abdominal ultrasound or CT, bone scintigraphy or FDG-PET-CT).
3. Bilateral synchronous or metachronous invasive breast cancer (in situ carcinoma of the contralateral breast is allowed)
4. Inflammatory breast cancer
5. Patients with a history of malignancy, other than invasive breast cancer, with the following exceptions:

   * Patients diagnosed, treated and disease-free for at least 5 years and deemed by the investigator to be at low risk for recurrence of that malignancy are eligible.
   * Patients with the following malignancies are eligible, even if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast; cervical cancer in situ; thyroid cancer in situ; non-metastatic, non-melanomatous skin cancers.
6. Previous treatment with palbociclib or any other CDK 4/6 inhibitors
7. Previous or planned chemotherapy or planned radiotherapy for the ipsilateral isolated locoregional recurrence (radiotherapy is allowed, but must be completed more than 2 weeks prior to randomization)
8. Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical disorder that would interfere with the patient's safety
9. Pregnant or lactating women; lactation has to stop before randomization
10. Patients with psychiatric illness/social situations that would limit compliance with study requirements
11. Contraindications or known hypersensitivity to the palbociclib or excipients
12. History of extensive disseminated/bilateral or known presence of interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and pulmonary fibrosis. A history of prior radiation pneumonitis is not considered an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Duration of invasive disease free survival of all randomized participants. | Assessed from the date treatment starts until the date of first documented invasive local, regional or distant recurrence, a second invasive cancer or death, or until approximately 4 years after treatment stops.
  Defined as the time from randomization until first appearance of invasive local, regional or distant recurrence (including invasive ipsilateral breast tumour recurrence), invasive contralateral breast cancer, a second (non-breast) invasive cancer, or death from any cause. The sites of first invasive disease events will be compared between treatment groups using a stratified log-rank test and will be tabulated.

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events. | Adverse events will be collected from the date consent is signed, and during treatment until 30-60 days after treatment stops.
  Adverse events, defined as any untoward medical occurrence, will be collected using CTCAE v5. All grades for targeted adverse events will be collected and all grades ≥3 for non-targeted adverse events. The maximum grade of each targeted adverse event during the protocol treatment phase will be determined, the frequencies summarized and tabulated according to grade and treatment assignment.
Duration of breast cancer free interval of all randomized participants. | Assessed from the date of randomization until the date of first documented breast cancer recurrence, or until approximately 4 years after treatment stops.
  Defined as the time from randomization until the date of first documented appearance of invasive local, regional or distant recurrence (including ipsilateral tumour recurrence), or invasive contralateral breast cancer.
Duration of distant recurrence free interval of all randomized participants. | Assessed from the date of randomization until the date of first documented distant disease progression, or until approximately 4 years after treatment stops.
  Defined as the time from randomization until the date of first documented distant recurrence of breast cancer.
Duration of overall survival of all randomized participants. | Assessed from the date of randomization until approximately 4 years after treatment stops, or until the date of death from any cause.
  Defined as the time from randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzone, MD, Study Chair — European Institute of Oncology
Locations (53):
- Austria (4):
  - Medizinische Universität Graz (MUG), Graz
  - Medizinische Universität Innsbruck - Univ.-Klinik f. Frauenheilkunde, Innsbruck
  - Uniklinikum Salzburg, Salzburg
  - MUW - Universitätsklinik für Innere Medizin, Vienna
- France (14):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Francois Baclesse, Caen
  - Cêntre Hospitaler de Cholet, Cholet
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Groupe hospitalier de Bretagne Sud, Hôpital du Scorff, Lorient
  - Centre Leon Berard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- National Institute of Oncology, Budapest, Hungary
- Italy (10):
  - Cro Irccs, Aviano
  - ASST Papa Giovanni XXIII, Bergamo
  - PO Antonio Perrino Brindisi, Brindisi
  - Istituto scientifico Romagnolo per lo studio e la cura, Meldola
  - Istituto Europeo di Oncologia, Milan
  - AOU Maggiore Della Carita, University of Eastern Piedmont, Novara
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Ospedale S. Stefano, Prato
  - U.O. Oncologia, Ospedale Infermi, Rimini
- Spain (14):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario de La Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d´Hebrón, Barcelona
  - Instituto Catalan de Oncologia L´Hospitalet, Barcelona
  - Hospital de Basurto, Bilbao
  - Institut Català d´Oncología (ICO), Girona
  - Hospital Universitario 12 de Octubre, Madrid
  - HU Ramón y Cajal, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Virgen de la Macarena, Seville
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (10):
  - Kantonsspital Baden, Baden
  - Brustzentrum Basel Bethesda Spital, Basel
  - Inselspital Bern, Bern
  - Centre du Sein Fribourg, Fribourg
  - Fondazione Oncologia Lago Maggiore, Locarno
  - Kouros Moccia Oncologia, Locarno
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Winterthur, Winterthur
  - BZ Bethanien, Zurich
  - Brust-Zentrum AG Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson SJ, Wapnir I, Dignam JJ, Fisher B, Mamounas EP, Jeong JH, Geyer CE Jr, Wickerham DL, Costantino JP, Wolmark N. Prognosis after ipsilateral breast tumor recurrence and locoregional recurrences in patients treated by breast-conserving therapy in five National Surgical Adjuvant Breast and Bowel Project protocols of node-negative breast cancer. J Clin Oncol. 2009 May 20;27(15):2466-73. doi: 10.1200/JCO.2008.19.8424. Epub 2009 Apr 6. PMID 19349544
- [Background] Wapnir IL, Aebi S, Geyer CE, Zahrieh D, Gelber RD, Anderson SJ, Robidoux A, Bernhard J, Maibach R, Castiglione-Gertsch M, Coates AS, Piccart MJ, Clemons MJ, Costantino JP, Wolmark N; IBCSG; BIG; NSABP. A randomized clinical trial of adjuvant chemotherapy for radically resected locoregional relapse of breast cancer: IBCSG 27-02, BIG 1-02, and NSABP B-37. Clin Breast Cancer. 2008 Jun;8(3):287-92. doi: 10.3816/CBC.2008.n.035. PMID 18650162
- [Background] Borner M, Bacchi M, Goldhirsch A, Greiner R, Harder F, Castiglione M, Jungi WF, Thurlimann B, Cavalli F, Obrecht JP, et al. First isolated locoregional recurrence following mastectomy for breast cancer: results of a phase III multicenter study comparing systemic treatment with observation after excision and radiation. Swiss Group for Clinical Cancer Research. J Clin Oncol. 1994 Oct;12(10):2071-7. doi: 10.1200/JCO.1994.12.10.2071. PMID 7931476
- [Background] Aebi S, Gelber S, Anderson SJ, Lang I, Robidoux A, Martin M, Nortier JW, Paterson AH, Rimawi MF, Canada JM, Thurlimann B, Murray E, Mamounas EP, Geyer CE Jr, Price KN, Coates AS, Gelber RD, Rastogi P, Wolmark N, Wapnir IL; CALOR investigators. Chemotherapy for isolated locoregional recurrence of breast cancer (CALOR): a randomised trial. Lancet Oncol. 2014 Feb;15(2):156-63. doi: 10.1016/S1470-2045(13)70589-8. Epub 2014 Jan 16. PMID 24439313
- [Background] Wapnir IL, Price KN, Anderson SJ, Robidoux A, Martin M, Nortier JWR, Paterson AHG, Rimawi MF, Lang I, Baena-Canada JM, Thurlimann B, Mamounas EP, Geyer CE Jr, Gelber S, Coates AS, Gelber RD, Rastogi P, Regan MM, Wolmark N, Aebi S; International Breast Cancer Study Group; NRG Oncology, GEICAM Spanish Breast Cancer Group, BOOG Dutch Breast Cancer Trialists' Group; Breast International Group. Efficacy of Chemotherapy for ER-Negative and ER-Positive Isolated Locoregional Recurrence of Breast Cancer: Final Analysis of the CALOR Trial. J Clin Oncol. 2018 Apr 10;36(11):1073-1079. doi: 10.1200/JCO.2017.76.5719. Epub 2018 Feb 14. PMID 29443653
- [Background] Migliaccio I, Di Leo A, Malorni L. Cyclin-dependent kinase 4/6 inhibitors in breast cancer therapy. Curr Opin Oncol. 2014 Nov;26(6):568-75. doi: 10.1097/CCO.0000000000000129. PMID 25188473
- [Background] Wardell SE, Ellis MJ, Alley HM, Eisele K, VanArsdale T, Dann SG, Arndt KT, Primeau T, Griffin E, Shao J, Crowder R, Lai JP, Norris JD, McDonnell DP, Li S. Efficacy of SERD/SERM Hybrid-CDK4/6 Inhibitor Combinations in Models of Endocrine Therapy-Resistant Breast Cancer. Clin Cancer Res. 2015 Nov 15;21(22):5121-5130. doi: 10.1158/1078-0432.CCR-15-0360. Epub 2015 May 19. PMID 25991817
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] Turner NC, Huang Bartlett C, Cristofanilli M. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Oct 22;373(17):1672-3. doi: 10.1056/NEJMc1510345. No abstract available. PMID 26488700